CLINICAL TRIAL: NCT00097500
Title: A Phase 3, Randomized, Open Label, Comparator-Controlled, Parallel Group, Multicenter Study to Compare the Effects of Exenatide and Insulin Glargine on Beta Cell Function and Cardiovascular Risk Markers in Subjects With Type 2 Diabetes Treated With Metformin Who Have Not Achieved Target HbA1c
Brief Title: Effects of Exenatide and Insulin Glargine in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2993-114
Record Dates: First submitted 2004-11-24; First posted 2004-11-25 (Estimated); Results first posted 2011-01-10 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; exenatide; exendin-4; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Insulin Glargine; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide Arm (Experimental): Exenatide and Metformin
  Interventions: Drug: exenatide; Drug: Metformin
- Insulin Glargine Arm (Active Comparator): Insulin Glargine and Metformin
  Interventions: Drug: Insulin glargine; Drug: Metformin

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, titrated up to a maximum of 20mcg three times a day in order to meet defined blood glucose targets
  Other Names: Byetta
  Arms: Exenatide Arm
Drug: Insulin glargine — subcutaneous injection, once a day, titrated as necessary in order to meet defined blood glucose targets
  Other Names: Lantus
  Arms: Insulin Glargine Arm
Drug: Metformin — Patients usual dosage

SUMMARY:
This Phase 3, open-label, multicenter study is designed to compare the effects of exenatide and insulin glargine (Lantus® injection) on beta-cell function in patients with type 2 diabetes mellitus using metformin.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes, but otherwise healthy
* HbA1c between 6.6% and 9.5%, inclusive.
* Body mass index (BMI) of 25 kg/m2 to 40 kg/m2, inclusive.
* Treated with a stable dose of metformin for at least 2 months prior to screening.

Exclusion Criteria:

* Patients previously in a study using exenatide.
* Treated with oral anti-diabetic medications other than metformin within 2 months of screening (thiazolidinediones within 5 months of screening).
* Treated with insulin within 3 months of screening.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2004-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Research and Development, MD, Study Director — Amylin Pharmaceuticals, LLC.
Locations (3):
- Research Site, Helsinki, Finland
- Research Site, Amsterdam, Netherlands
- Research Site, Gothenburg, Sweden

REFERENCES:
- [Result] Bunck MC, Diamant M, Corner A, Eliasson B, Malloy JL, Shaginian RM, Deng W, Kendall DM, Taskinen MR, Smith U, Yki-Jarvinen H, Heine RJ. One-year treatment with exenatide improves beta-cell function, compared with insulin glargine, in metformin-treated type 2 diabetic patients: a randomized, controlled trial. Diabetes Care. 2009 May;32(5):762-8. doi: 10.2337/dc08-1797. Epub 2009 Feb 5. PMID 19196887
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Muskiet MHA, Bunck MC, Heine RJ, Corner A, Yki-Jarvinen H, Eliasson B, Joles JA, Diamant M, Tonneijck L, van Raalte DH. Exenatide twice-daily does not affect renal function or albuminuria compared to titrated insulin glargine in patients with type 2 diabetes mellitus: A post-hoc analysis of a 52-week randomised trial. Diabetes Res Clin Pract. 2019 Jul;153:14-22. doi: 10.1016/j.diabres.2019.05.001. Epub 2019 May 9. PMID 31078666
- [Derived] Bunck MC, Corner A, Eliasson B, Heine RJ, Shaginian RM, Taskinen MR, Smith U, Yki-Jarvinen H, Diamant M. Effects of exenatide on measures of beta-cell function after 3 years in metformin-treated patients with type 2 diabetes. Diabetes Care. 2011 Sep;34(9):2041-7. doi: 10.2337/dc11-0291. PMID 21868779
- [Derived] Bunck MC, Corner A, Eliasson B, Heine RJ, Shaginian RM, Wu Y, Yan P, Smith U, Yki-Jarvinen H, Diamant M, Taskinen MR. One-year treatment with exenatide vs. insulin glargine: effects on postprandial glycemia, lipid profiles, and oxidative stress. Atherosclerosis. 2010 Sep;212(1):223-9. doi: 10.1016/j.atherosclerosis.2010.04.024. Epub 2010 Apr 29. PMID 20494360

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Arm: 5 mcg twice a day for 4 weeks, followed by 10 mcg twice a day for 8 weeks. After 12 weeks, exenatide is titrated (up to a maximum of 20 mcg three times a day) based on periodic glycosylated hemoglobin (HbA1c) measurements and tolerability.
- Insulin Glargine Arm: Dosing starts at 10 IU/day, and is then titrated, based on daily fasting blood glucose measurements.
Period: On-drug Period (Week 0 to Week 52)
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Started | 36 | 33
Completed | 30 (Subjects experiencing loss of glucose control after Week 52 are considered to have completed study.) | 30 (Subjects experiencing loss of glucose control after Week 52 are considered to have completed study.)
Not Completed | 6 | 3
Not completed — Withdrawal of consent | 1 | 1
Not completed — Adverse Event | 5 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Off-drug Period (Week 52 to Week 64)
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Started | 30 (Exenatide is discontinued, metformin is continued) | 30 (Insulin Glargine is discontinued, metformin is continued)
Completed | 25 | 26
Not Completed | 5 | 4
Not completed — Withdrawal of consent | 2 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Loss of glucose control | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Arm | Insulin Glargine Arm | Total
Number analyzed (Participants) | 36 | 33 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (8.4) | 58.3 (7.3) | 58.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 23 | 22 | 45
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.87 (4.15) | 30.13 (3.49) | 30.52 (3.84)
Body weight [Mean (Standard Deviation); unit: kg] | 90.56 (12.66) | 92.39 (13.56) | 91.44 (13.03)
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage] | 7.58 (0.89) | 7.41 (0.81) | 7.50 (0.85)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 5.72 (4.70) | 3.97 (3.62) | 4.88 (4.28)

OUTCOME MEASURES:

1. Primary Outcome: Beta-cell Function After 52 Weeks of Therapy
Description: Treatment effect on beta-cell function as measured by the ratio of Week 52 arginine-stimulated insulin secretion during a hyperglycemic clamp(specifically, the incremental AUC of insulin with respect to basal value over a 10 min period [i.e., clamp time 290 min to 300 min]) to that at baseline (i.e., the ratio is calculated as arginine-stimulated insulin secretion at week 52 divided by arginine-stimulated insulin secretion at baseline [week -2]).
Time Frame: Baseline (week -2) and 52 weeks
Population: Evaluable population
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 30 | 30
ratio | 2.89 (0.27) | 1.15 (0.11)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p = 0.0001, ANCOVA

2. Secondary Outcome: Beta-cell Function 4 Weeks After Cessation of Therapy
Description: Treatment effect on beta-cell function as measured by the ratio of Week 56 arginine-stimulated insulin secretion during a hyperglycemic clamp(specifically, the incremental AUC of insulin with respect to basal value over a 10 min period [i.e., clamp time 290 min to 300 min]) to that at baseline (i.e., the ratio is calculated as arginine-stimulated insulin secretion at week 56 divided by arginine-stimulated insulin secretion at baseline [week -2]).
Time Frame: Baseline (week -2) and 56 weeks
Population: Evaluable population
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 30 | 30
ratio | 1.02 (0.06) | 1.08 (0.07)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p = 0.4185, ANCOVA

3. Secondary Outcome: Change in First Phase C-peptide Release
Description: Ratio of first phase C-peptide response to glucose at 52 weeks (end of on-drug period) and 56 weeks (during off-drug period) compared to first phase C-peptide response to glucose at baseline (i.e., C-peptide response to glucose at week 52 or week 56 divided by C-peptide response to glucose at baseline [week -2]). C-peptide is measured as a surrogate marker of insulin secretion. First phase C-peptide/insulin release is measured during the first ten minutes of glucose infusion during a hyperglycemic clamp procedure.
Time Frame: baseline (week -2), 52 weeks, and 56 weeks
Population: Evaluable population. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 29 | 30
ratio
  52 weeks | 1.72 (0.11) | 1.13 (0.07)
  56 weeks | 0.95 (0.05) | 1.06 (0.06)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Statistical analysis at week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Exenatide Arm vs Insulin Glargine Arm; Statistical analysis at week 56; Test type: Superiority or Other; p = 0.1188, ANCOVA

4. Secondary Outcome: Change in Second Phase C-peptide Release
Description: Ratio of second phase C-peptide response to glucose at 52 weeks (end of on-drug period) and 56 weeks (during off-drug period) compared to second phase C-peptide response to glucose at baseline (i.e., C-peptide response to glucose at week 52 or week 56 divided by C-peptide response to glucose at baseline [week -2]). C-peptide is measured as a surrogate marker of insulin secretion. Second phase C-peptide/insulin release is measured from time=10 minutes to time=80 minutes of glucose infusion during a hyperglycemic clamp procedure.
Time Frame: baseline (-2 weeks), 52 weeks, and 56 weeks
Population: Evaluable population. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 30 | 30
ratio
  52 weeks | 2.88 (0.18) | 1.01 (0.07)
  56 weeks | 1.00 (0.05) | 1.08 (0.06)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Statistical analysis at week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA
Statistical Analysis 2: Comparison: Exenatide Arm vs Insulin Glargine Arm; Statistical analysis at week 56; Test type: Superiority or Other; p = 0.1996, ANCOVA

5. Secondary Outcome: Change in Glycosylated Hemoglobin (HbA1c)
Description: Change in HbA1c from week 0 to week 52 (i.e., HbA1c at week 52 minus HbA1c at week 0).
Time Frame: Week 0 and week 52
Population: Intent to treat population. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 36 | 33
percent | -0.97 (0.14) | -0.87 (0.15)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p = 0.5522, ANCOVA

6. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose from week 0 to week 52 (i.e., fasting plasma glucose at week 52 minus fasting plasma glucose at week 0).
Time Frame: 0 weeks and 52 weeks
Population: Intent to treat population. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 36 | 33
mmol/L | -1.53 (0.25) | -3.10 (0.27)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p < 0.0001, ANCOVA

7. Secondary Outcome: Seven Point Self Monitored Blood Glucose (SMBG) Measurements
Description: SMBG measured at 7 time points (before and after breakfast, before and after lunch, before and after dinner, at bedtime).
Time Frame: 0 weeks and 52 weeks
Population: Intent to treat population.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 36 | 33
mmol/L
  Pre-breakfast measurement (week 0) | 8.92 (1.80) | 8.38 (1.91)
  Pre-breakfast measurement (week 52) | 7.27 (1.63) | 5.63 (0.85)
  2-hour post-breakfast measurement (week 0) | 11.00 (2.58) | 11.17 (3.30)
  2-hour post-breakfast measurement (week 52) | 6.98 (2.42) | 7.53 (2.16)
  Pre-lunch measurement (week 0) | 8.14 (2.25) | 8.54 (2.51)
  Pre-lunch measurement (week 52) | 6.52 (1.52) | 6.24 (1.66)
  2-hour post-lunch measurement (week 0) | 9.90 (2.54) | 10.52 (2.96)
  2-hour post-lunch measurement (week 52) | 7.97 (2.01) | 8.15 (1.77)
  Pre-dinner measurement (week 0) | 8.38 (2.40) | 8.07 (2.48)
  Pre-dinner measurement (week 52) | 7.53 (2.63) | 6.98 (2.04)
  2-hour post-dinner measurement (week 0) | 10.42 (2.42) | 10.26 (2.82)
  2-hour post-dinner measurement (week 52) | 6.98 (2.25) | 8.81 (2.03)
  Bedtime measurement (week 0) | 9.76 (2.44) | 9.85 (3.09)
  Bedtime measurement (week 52) | 7.61 (2.11) | 8.03 (2.82)

8. Secondary Outcome: Change in Body Weight
Description: Change in body weight from week 0 to week 52 (i.e., body weight at week 52 minus body weight at week 0).
Time Frame: 0 weeks and 52 weeks
Population: Intent to treat population. Last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 36 | 33
kg | -3.80 (0.87) | 0.75 (0.95)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p < 0.0001, ANCOVA

9. Secondary Outcome: M-value at Baseline, Week 52 and Week 56
Description: M-value at baseline (week -2), week 52 (end of on-drug period), and week 56 (during off-drug period). Insulin sensitivity was assessed during the euglycemic/hyperglycemic clamp test at baseline (week -2), week 52, and week 56. Insulin-mediated glucose uptake (M-value) was calculated as the mean glucose requirement during the 90-120 minute interval of the clamp.
Time Frame: baseline (week -2), 52 weeks, and 56 weeks
Population: Evaluable population.
Measure: Mean (Standard Error); unit: mg/min/kg
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 30 | 30
mg/min/kg
  baseline (week -2) | 2.24 (0.39) | 2.79 (0.26)
  week 52 | 3.18 (0.42) | 3.85 (0.32)
  week 56 | 3.19 (0.44) | 2.81 (0.29)

ADVERSE EVENTS:
Time Frame: Total reporting period for adverse events is 64 weeks: a 52-week on-drug period followed by a 12-week off-drug period.
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Serious Adverse Events (participants affected / at risk) | 3/36 | 1/33
Other Adverse Events (participants affected / at risk) | 32/36 | 31/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Arm (N=36) | Insulin Glargine Arm (N=33)
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Thrombophlebitis Superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Arm (N=36) | Insulin Glargine Arm (N=33)
Anemia (Blood and lymphatic system disorders) | 1 | 4
Abdominal Distension (Gastrointestinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 5 | 2
Flatulence (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 18 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Injection Site Rash (General disorders) | 3 | 0
Edema Peripheral (General disorders) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 4
Influenza (Infections and infestations) | 5 | 9
Laryngitis (Infections and infestations) | 2 | 1
Tooth Infection (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 3 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 0
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 6 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days